CLINICAL TRIAL: NCT05677308
Title: LYNPARZA Tablets 100mg, 150mg General Drug Use-results Study in Patients With BRCA Mutated HER2 Negative High Recurrent Risk Breast Cancer in the Adjuvant Setting
Brief Title: LYNPARZA Breast Cancer in the Adjuvant Setting Japan Post-Marketing Surveillance (PMS)
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D081CC00012
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To evaluate the frequency of bone marrow suppression Adverse Drug Reactions (ADRs) in patients with BRCA mutated HER2 negative high recurrent risk breast cancer treated with LYNPARZA for adjuvant treatment in the actual post-marketing use.

DETAILED DESCRIPTION:
To evaluate the frequency of bone marrow suppression Adverse Drug Reactions (ADRs) in patients with BRCA mutated HER2 negative high recurrent risk breast cancer treated with LYNPARZA for adjuvant treatment in the actual post-marketing use.

This investigation will be conducted for application for re-examination specified in Article 14-4 of the Pharmaceutical Affairs Law.

ELIGIBILITY:
Inclusion Criteria:

* The patients who started treatment with LYNPARZA for the first time for the approved indication "Adjuvant treatment for patients with BRCA-mutated HER2 negative high recurrent risk breast cancer"

Exclusion Criteria:

* Patients who have no treatment history with LYNPARZA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who started treatment with LYNPARZA for "Adjuvant treatment for patients with BRCA-mutated HER2 negative high recurrent risk breast cancer"
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of bone marrow suppression | from baseline to 1year

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (39):
- Japan (39):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home